CLINICAL TRIAL: NCT01621451
Title: Does Early Re-administration of Aspirin/Clopidogrel Increase the Risk of Bleeding From Artificial Ulcer After EMR or ESD?
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Asan Medical Center (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Hwoon-Yong Jung, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PZ-1001-403-NS
Record Dates: First submitted 2012-06-13; First posted 2012-06-18 (Estimated); Last update posted 2012-11-22 (Estimated); Status verified 2012-11

CONDITIONS: Early Gastric Cancer; Gastric Dysplasia
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- immediate (Active Comparator): Patients who receive pantoprazole plus aspirin and/or clopidogrel within 3~4 days after EMR/ESD
  Interventions: Drug: aspirin and/or clopidogrel
- 2 weeks (Active Comparator): Patients who receive pantoprazole plus aspirin and/or clopidogrel at 2 weeks after EMR/ESD
  Interventions: Drug: aspirin and/or clopidogrel

INTERVENTIONS:
Drug: aspirin and/or clopidogrel — Patients who have taken aspirin and/or clopidogrel and are found to have early gastric cancer or gastric premalignant lesions including adenoma and dysplasia by upper endoscopy will be stopped aspirin and/or clopidogrel for 7 days before EMR/ESD. In immediate group, the patient will receive oral proton pump inhibitor (pantoprazole 40mg per day) for 4 weeks after EMR/ESD to treat their post-EMR/ESD ulcer.
  Arms: immediate
Drug: aspirin and/or clopidogrel — Patients who have taken aspirin and/or clopidogrel and are found to have early gastric cancer or gastric premalignant lesions including adenoma and dysplasia by upper endoscopy will be stopped aspirin and/or clopidogrel for 7 days before EMR/ESD.
  In 2 weeks group, the patient will receive oral proton pump inhibitor (pantoprazole 40mg per day) for 4 weeks after EMR/ESD to treat their post-EMR/ESD ulcer.
  Arms: 2 weeks

SUMMARY:
Aspirin and/or clopidogrel users are increasing due to increased prevalence of cardiovascular or cerebrovascular disease with an aging society in Korea. Also, the patients having endoscopic mucosal resection (EMR) or endoscopic submucosal dissection (ESD) for early gastric cancer or gastric premalignant lesions including adenoma and dysplasia are increasing among aspirin and/or clopidogrel users. Practically, aspirin or clopidogrel is recommended to be stopped for 5~14 days before EMR or ESD because bleeding risk during or after procedure. And it is recommended to restart of aspirin and/or clopidogrel as soon as possible if immediate bleeding during or after the procedure is not occurred in consideration of thromboembolic risk. However, early restarting of aspirin and/or clopidogrel raise the risk of delayed bleeding and the risk of complications associated with delayed ulcer healing. Although it is important to determine the timing of restarting aspirin and/or clopidogrel in consideration of complications of post-EMR/ESD ulcer and thromboembolic risk, there is no definite guideline about the timing of restarting aspirin and/or clopidogrel.

This study is aimed to determine the timing of restarting aspirin and/or clopidogrel for the patients having EMR or ESD among aspirin and/or clopidogrel users. The investigators planned to compare the delayed bleeding rate and ulcer healing rate in patients with post-EMR/ESD ulcer when take proton pump inhibitor (pantoprazole 40 mg per day) between the patients restarting aspirin and/or clopidogrel within 3~4 days after the procedure and the patients restarting aspirin and/or clopidogrel 2 weeks after the procedure during 4 weeks. The primary endpoint is delayed ulcer bleeding rate at 4 weeks after EMR/ESD. The secondary end point is ulcer healing rate within 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have taken aspirin and/or clopidogrel for cardiovascular and/or cerebrovascular disease and are found to have early gastric cancer or premalignant lesions including adenoma and dysplasia by upper endoscopy.

Exclusion Criteria:

* Patients with known coagulopathy or abnormal coagulation tests (prothrombin time, partial thromboplastin time and platelet count)
* Patients receiving other antithrombotic, anticoagulant drugs
* Patients needing continuation of nonsteroidal anti-inflammatory drugs, cyclooxygenase-2 (COX-2) inhibitors, or steroid after EMR/ESD
* Patient with recent percutaneous coronary intervention (placement of drug eluting coronary artery stent within 12 months, bare metal coronary artery stents within 1 month)
* Patient's age > 80 year-old or < 18 year-old
* Patient with severe cardiovascular, pulmonary, hepatic, or renal disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2012-06; Primary Completion 2014-05 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
delayed ulcer bleeding | 4 weeks

SECONDARY OUTCOMES:
ulcer healing rate | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hwoon-Yong Jung, professor, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea